CLINICAL TRIAL: NCT07387900
Title: Evaluation of the Chemo-preventive Effect of Combined Topical and Systemic Metformin on Oral Leukoplakia: A Randomized Clinical Trial
Brief Title: Evaluation of the Chemo-preventive Effect of Combined Topical and Systemic Metformin on Oral Leukoplakia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Refaat Elmohamady Soliman Ghanem, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OMED 3.7.2
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Oral Leukoplakia
Keywords: Oral Leukoplakia; Metformin
MeSH Terms: conditions — Leukoplakia, Oral | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical and systemic metformin (Experimental)
  Interventions: Drug: Metformin Hydrochloride
- Topical and systemic Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin Hydrochloride — 10% oral gel and 500mg tablet
  Arms: Topical and systemic metformin
Drug: Placebo — Placebo Gel and 500mg Placebo tablet
  Arms: Topical and systemic Placebo

SUMMARY:
There is no consensus on treatment of leukoplakia but surgical excision is the preferred choice if suitable in size, which does not prevent clinical recurrence and malignant transformation. Chemoprevention is a new direction in the management of OL using various topical and systemic agents such as; vitamin A, lycopene, celecoxib, green tea extract, and metformin.

While metformin cannot realistically be used as cancer mono-therapy, it can be used as an adjunct and can have a more promising effect on lesions that have yet to undergo malignant transformation. Thus, the aim of this study is to investigate the efficacy of combined chemo-preventive effect of topical and systemic Metformin on oral leukoplakia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 21 years.
* Patients clinically diagnosed and histologically confirmed as having oral Leukoplakia.
* Lesions with mild to moderate degree of dysplasia.
* Patients who agree to sign a written consent after understanding the nature of the study.

Exclusion Criteria:

* Patients with lesions showing sever degree of dysplasia.
* Patients who have cardiovascular, lung, Renal, Liver diseases
* Patients on metformin therapy (eg: Diabetes Mellitus, PCOS, …etc.)
* Patients on H2 blocker & proton pump inhibitors therapy as Ranitidine (affects metformin absorption and clearance)
* Those with allergy or sensitivity to Metformin therapy or having any contraindication for their use.
* Patients on Retinoid, green tea supplements or another natural products therapy
* Patients with other accompanying oral lesions
* Pregnant or Lactating females

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in lesion size | over 6 months
  the lesion will be measured in size by periodontal probe bi-dimensionally in mms

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt